CLINICAL TRIAL: NCT04572061
Title: Emergency Coronary Artery Bypass Graft in Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Saud Al Babtain Cardiac Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SBCC-2017-04
Record Dates: First submitted 2020-06-14; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute Myocardial Infarction
Keywords: CABG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study investigating the early outcome of emergency CABG post MI in patients who were operated at Saud Al Babtain Cardiac Center.

DETAILED DESCRIPTION:
A retrospective study of surgical patients who underwent Coronary Artery Bypass Graft for Acute Myocardial Infarction between December 2013 and February 2018 determining outcomes on morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post cardiogenic shock who underwent CABG
* =/> 17 years old

Exclusion Criteria:

* Patients other than post cardiogenic shock who underwent CABG or any cardiac surgeries
* <17 years old

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients admitted at Saud Al Babtain Cardiac Center with post cardiogenic shock who underwent CABG.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
STEMI and Emergency CABG | 1 year
  Evaluate patients the early outcome of emergency CABG post MI.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Attiea, MD, Principal Investigator — Saud Al Babtain Cardiac Center
Locations (1):
- Saud Al Babtain Cardiac Center, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided